CLINICAL TRIAL: NCT02954510
Title: Ferumoxytol-enhanced Magnetic Resonance Imaging for the Interpretation of Vascular Defects
Brief Title: Ferumoxytol-enhanced Magnetic Resonance Imaging
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Michael Siedlecki, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P000250
Record Dates: First submitted 2016-01-12; First posted 2016-11-03 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Intervention Model Description: case control
Masking Description: Experts evaluating ferumoxytol-enhanced magnetic resonance imaging will be masked to the results of other invasive and non-invasive cardiac testing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Single arm utilizing ferumoxytol
  Interventions: Drug: ferumoxytol

INTERVENTIONS:
Drug: ferumoxytol — ferumoxytol will assess patency of coronary arteries
  Other Names: feraheme

SUMMARY:
There are no current alternatives to diagnostic contrast-requiring imaging for patients with an eGFR <30mL/min due to the association of gadolinium-based imaging modalities to nephrogenic systemic fibrosis and iodinated contrast-induced kidney injury. Ferumoxytol-enhanced imaging may offer an alternative approach.

DETAILED DESCRIPTION:
This is a case control study which will assess the resolution by which the coronary arteries can be visualized using ferumoxytol-enhanced cardiac magnetic resonance angiography (fcMRA) in patients with prior regional cardiac ischemia localized by stress-induced echocardiography. Resolution will be compared to invasive coronary arteriography completed in all patients that will be analyzed at the end of the study.

Masked experts will interpret fcMRA images to determine if coronary stenosis is present or absent. By strict definitions, this is a single-arm study. However comparison will be made between fcMRA and invasive coronary arteriography performed in each patient. With a prevalence of disease of approximately 0.35 in the study population, it is anticipated that both sensitivity and specificity of fcMRA to identify the absence of coronary artery stenosis can be calculated.

We anticipate a population size of 70 will be needed to adequately study the primary outcome due to potential confounders, including racial and sex differences which may exist (see below), which are known to exist in a population with significant renal and possible cardiac disease to determine if fcMRA is differs in its ability to exclude greater than or equal to 50 percent stenosis in a single coronary artery compared to dobutamine stress echocardiography (DSE). This is based on prevalence of disease of 0.35. Non-invasive cardiac stress testing in those with eGFR <30ml/min/1.73m2 is estimated to have a sensitivity of 0.81 (CI 0.57-0.94) and specificity of 0.83 (CI 0.62-0.95) to identify coronary epicardial lesion of greater than 70 percent. The sensitivity of non-invasive non-intraluminal testing is anticipated to be 0.60 when patients with myocardial scar are enrolled. We anticipate that 50 percent of patients with a positive DSE will have evidence of myocardial scar. Predicted sensitivity of fcMRA will likely be increased compared to referenced estimates because true positives will be defined by stenosis greater than or equal to 50 percent. Based on a prevalence of 0.35, we anticipate DSE will yield 24 true positives, 25 true negatives, 7 false positives, and 14 false negatives resulting in sensitivity of 0.63 and specificity of 0.78. To achieve study power that will allow for the null hypothesis to be ignored, in as study size of 70, fcMRA must yield at least 28 true positives and 27 true negatives allowing for 5 false positives and 10 false negatives resulting in sensitivity of 0.737 and specificity of 0.843. To account for drop-out and incomplete data collection in 50 percent of patients approached, recruitment of 140 patients will be needed. The drop-out rate from recruitment to enrollment approximates the fcMRA study experience at the Brigham and Women's Hosptial in 2017.

Racial/sex subgroup analysis will involve testing in whites vs. non-whites and males vs. females. Prevalence of 0.35 will again be assumed. Previously, 45 percent of patients enrolled were of non-white racial origin. An additional 85 patients would be necessary to demonstrate a difference between fcMRA and DSE when comparing sensitivity and specificity as above, therefore this will be considered an exploratory analysis.

Using the Partners Healthcare System Research Patient Data Registry (RPDR) all patients in calendar year 2017 were identified with a diagnosis of chronic kidney disease stage 4-5D and who underwent a left heart cardiac catheterization at either Brigham and Women's Hospital or Massachusetts General Hospital (MGH). "chronic kidney disease stage 4", "chronic kidney disease stage 5", and "left heart catheterization", and "abnormal echocardiogram" were used as mesh terms resulting in 68 patients. 108 patients utilizing hemodialysis or peritoneal dialysis completed ICA. 35 patients not yet requiring renal replacement therapy completed ICA in the same time period. Separately, clinical practices at the Brigham and Women's Hospital kidney transplant center in calendar year 2017 were reviewed. 207 patients underwent non-invasive cardiac stress testing and 16 patients underwent ICA. All patients that underwent arteriography had prior non--invasive cardiac stress testing. Surveying both the inpatient and outpatient settings a total of 159 patients were identified in the Partners Healthcare System that would have qualified for the proposed study.

ELIGIBILITY:
Both female and male participants are being studied aged 18-85 years old with an estimated glomerular filtration rate (eGFR) of less than 30ml/min/1.73 meters squared. Patients will have undergone cardiac screening tests that warrant further evaluation. Patients will be excluded with an eGFR >30ml/min/1.73 meters squared.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-27 (Estimated)

PRIMARY OUTCOMES:
Detect the absence of ≥50% stenosis in the coronary artery tree | 48 months
  This outcome derives from the central hypothesis which states that coronary artery disease can more effectively be excluded in patients with severe chronic kidney disease using ferumoxtyol enhanced cardiac magnetic resonance angiography (fcMRA) rather than non-invasive cardiac testing combined with ICA. The presence or absence of a single 50% stenosis in the region of interest (measured as described above) will be dichotomized (0=absent/ 1= present) from each of the two measures, fcMRA and invasive coronary arteriography

SECONDARY OUTCOMES:
Detect stenosis in proximal and distal segments of the coronary artery tree | 48 months
  The purpose of this secondary outcome is to determine the sensitivity and specificity of fcMRA to detect the absence of lesions exhibiting ≥50% stenosis compared to ICA in proximal and distal arterial segments
Compare ferumoxtyol enhanced magnetic resonance angiography with stress echocardiography | 48 months
  The purpose of this secondary outcome is to determine the contrast and estimate the similarity between fcMRA, dobutamine stress echocardgiography testing with the gold standard of ICA

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study de-identified data will be made available. according to guidelines described by the Biological Specimen and Data Repository Information Coordinating Center. The structure will abide by the National Heart Lung Blood Institute Policy for Data Sharing from Clinical Trials and Epidemiological Studies.
Time Frame: Within one year of the conclusion of the study. Data will be available for at least seven years.

REFERENCES:
- [Derived] Chin MS, Steigner M, Yin W, Kwong RY, Siedlecki AM. Intraluminal Assessment of Coronary Arteries With Ferumoxytol-Enhanced Magnetic Resonance Angiography. JACC Cardiovasc Imaging. 2018 Mar;11(3):505-508. doi: 10.1016/j.jcmg.2017.10.017. Epub 2017 Dec 13. No abstract available. PMID 29248659